CLINICAL TRIAL: NCT01971879
Title: Protection of Arteritic Patients by Remote Preconditioning
Acronym: PARADIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: AOI 2012-07
Record Dates: First submitted 2013-10-17; First posted 2013-10-29 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Obliterating Arteriopathy of the Lower Limbs
Keywords: Remote ischemic preconditioning; Obliterating Arteriopathy of the Lower Limbs

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Sham Comparator)
  Interventions: Procedure: Control
- Remote preconditioning (Active Comparator)
  Interventions: Procedure: Remote ischemic preconditioning

INTERVENTIONS:
Procedure: Remote ischemic preconditioning — A blood pressure cuff is placed on one arm and is inflated to 200mmHg during 5 minutes. During the following 5 minutes, the cuff is inflated at the same pressure on the contralateral arm. This sequence is repeated 3 times, that is to say 3 sequences of cuff inflation for 5 minutes on each arm followed by 5 minutes without inflation.
  The treadmill test starts 5 minutes after the end of the last deflation of the cuff.
  Arms: Remote preconditioning
Procedure: Control — A blood pressure cuff is placed on one arm and is inflated to 10mmHg during 5 minutes. During the following 5 minutes, the cuff is inflated at the same pressure on the contralateral arm. This sequence is repeated 3 times, that is to say 3 sequences of cuff inflation for 5 minutes on each arm followed by 5 minutes without inflation.
  The treadmill test starts 5 minutes after the end of the last deflation of the cuff.
  Arms: Control

SUMMARY:
Prospective, monocentric, randomised, double-blind study with 20 patients enrolled to be explored twice through a Cross-over strategy to determine whether remote preconditioning improves arteritic patients' ability to walk.

DETAILED DESCRIPTION:
Patients will be screened amongst arteritic patients who have undergone a positive treadmill test in Angers University Hospital, defined by a premature test stop caused by muscular pain associated to trans-cutaneous pressure of oxygen (TCPO2) drop.

After signing the informed consent, patients will take two treadmill tests in a week-span. According to randomization, patients will undergo the "remote preconditioning" procedure or the "control" procedure before the first treadmill test. The following week, in respect to a cross-over strategy patients will undergo the other procedure before the second treadmill test.

Only the study nurse will be advised of the procedure to do. Investigators will not be informed about the allocated procedure. Patients will not be informed about the procedure supposed to have a beneficial effect.

The treadmill test will be run according to a calibrated protocol. After a 2-minute stand-up resting period, the treadmill will progressively speed up to a 3.2km/h during one minute. This stage will be maintained with a 10% slope for 14 minutes. Then, the treadmill's slope and speed will increase progressively every minute according to a calibrated protocol. The test duration will be measured from the start of the walk to the patient's request to stop because of pain in the lower limbs.

TCPO2 will be measured before and during the test on the glutei and the legs. Tissue oxygenation on both lower limbs will be measured by Near Infra-Red Spectroscopy (NIRO-200NX system). Oxygen consumption will be analysed throughout the test.

A blood sample will be drawn just before the start of the test, that is 5 minutes after the end of the last cuff deflation. A second blood sample will be drawn 2 minutes after the patient's request to stop walking. These blood samples are composed of one 3ml tube to measure out blood lactate level, one 6ml ethylene diamine tetraacetic acid (EDTA) tube and a 5ml plain tube. These two last tubes will be centrifuged and subsampled to build up a bio-collection stored at the local Biological Resources Center.

ELIGIBILITY:
Inclusion Criteria:

* Positive treadmill test (maximum walking distance < 750m because of lower limbs muscular pain)
* Resting systolic pressure index < 0,9 (uni- or bilateral)
* Resting systolic blood pressure <200mmHg
* Written informed consent
* Affiliation to a Social Security scheme

Exclusion Criteria:

* Effort hypoxemia during the selection treadmill test
* Patient treated with metformin during the 7 days preceding the treadmill tests
* Person who is not affiliated to a Social Security scheme or benefiting from such a scheme
* Person in an exclusion period related to another biomedical study
* Patient refusal / patient not having provided written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-10; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Walking distance during the calibrated treadmill test | 1 week

SECONDARY OUTCOMES:
Tissue oxygenation measure by Near Infra-Red Spectroscopy during the test | 1 week
TCPO2 half-rise time measure after the test | 1 week
Measure of the deepness of TCPO2 drop | 1 week
Heart rate measured 1 min and 2 min after test stop/ resting heart rate before test | 1 week
Oxygen consumption analyse during the effort (VO2) | 1 week
Lactate blood level at the end of the test | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice PRUNIER, Professor, Study Director — University Hospital, Angers; Sylvain GRALL, Doctor, Principal Investigator — University Hospital, Angers
Locations (1):
- Service de Médecine du Sport, CHU d'Angers, Angers, France